CLINICAL TRIAL: NCT06689839
Title: A Prospective, Randomized, Multicenter, Single-blind Trial to Assess the Safety and Effectiveness of the Encompass F2 Cerebral Protection System Vs. Standard of Care (Unprotected or Sentinel® Cerebral Protection System) During Transfemoral Transcatheter Aortic Valve Replacement
Brief Title: Trial of the F2 Filter and Delivery System for Embolic Protection During TAVR
Acronym: SHIELD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EnCompass Technologies, Inc. (Industry)
Collaborators: Avania (Industry); Insight Medical Consulting (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ET03
Record Dates: First submitted 2024-11-01; First posted 2024-11-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis Treated With TAVI; Aortic Diseases
Keywords: Embolic Protection; Transcatheter Aortic Valve Replacement; TAVR; Aortic Valve Stenosis; Aortic Valve Diseases
MeSH Terms: conditions — Aortic Diseases; Aortic Valve Stenosis; Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 1:1 ratio to:
  * Transcatheter Aortic Valve Replacement (TF TAVR) with the F2 Cerebral Protection System (CPS) (treatment group) or
  * Transcatheter Aortic Valve Replacement (TF TAVR) with Standard of Care treatment (no embolic protection or use of the commercially available protection device, Sentinel System; control group)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- F2 Filter and Delivery System (Experimental): The F2 Cerebral Embolic Protection System will be used during your Transcatheter Aortic Valve Replacement procedure
  Interventions: Device: F2 Filter and Delivery System; Procedure: Transcatheter Aortic Valve Replacement (TAVR)
- Either the Sentinel Cerebral Protection System or no embolic protection device (Active Comparator): Either the Sentinel Cerebral Protection System or no embolic protection device will be used during your Transcatheter Aortic Valve Replacement procedure depending on the Standard of Care at the treating institution
  Interventions: Procedure: Transcatheter Aortic Valve Replacement (TAVR)

INTERVENTIONS:
Device: F2 Filter and Delivery System — Use of the F2 Filter and Delivery System in conjunction with a Transcatheter Aortic Valve Replacement (TAVR) procedure
  Arms: F2 Filter and Delivery System
Procedure: Transcatheter Aortic Valve Replacement (TAVR) — Transcatheter Aortic Valve Replacement (TAVR) with commercially available Transcatheter Aortic Valve Replacement (TAVR) device

SUMMARY:
The objective of this study is to compare the safety and effectiveness of the F2 Cerebral Protection System (CPS) to a standard of care control group in patients undergoing Transcatheter Aortic Valve Replacement (TF TAVR)

DETAILED DESCRIPTION:
The study is designed to demonstrate that the F2 Cerebral Protection System (CPS) performs in a consistent manner as the control group in terms of safety, and the F2 Cerebral Protection System (CPS) will be superior in performance when compared to the control group in terms of effectiveness in patients undergoing Transcatheter Aortic Valve Replacement (TF TAVR).

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 50 years.
* Patient meets the established criteria and indications for commercially available TAVR via transfemoral access and is scheduled to undergo TAVR per their treating physician.
* Patient is willing and able to comply with protocol-specified follow-up evaluations.
* Patient is able and willing to provide written informed consent.
* Patient meets all criteria for use of control device (Sentinel device, per IFU).

Key Exclusion Criteria:

General Exclusion Criteria:

* Patient requires an urgent or emergent TAVR procedure.
* Any interventional cardiovascular procedure performed within 30 days prior to TAVR procedure or planned within 30 days post-TAVR procedure.
* Diagnostic cardiac catheterization within 10 days prior to TAVR procedure.
* Evidence of an acute myocardial infarction within 3 months prior to TAVR procedure.
* Prior prosthetic heart valve in any position.
* Known intracardiac thrombus.
* Active infection or endocarditis.
* Patient is contraindicated for anti-platelet and/or anticoagulant therapy.
* Patient refuses blood transfusion.
* Renal insufficiency (creatinine > 2.5 mg/dL or GFR < 30) and/or renal replacement therapy at the time of screening.
* Patients with hepatic failure (Child-Pugh class C).
* Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 30%.
* Females who are pregnant or nursing or plan to become pregnant during their participation in the study.

Neurological Exclusion Criteria:

* Modified Rankin Scale (mRS) ≥ 2 at screening.
* Cerebrovascular event including TIA within 6 months of the procedure.
* Patient has active major psychiatric disease, known mental or physical illness or known history of substance abuse that may cause non-compliance with the protocol or confound the data interpretation.
* Patient has severe visual, auditory, or learning impairment.
* Patient has neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.

Magnetic Resonance Imaging Exclusion Criteria:

* Contraindications to MRI (participants with MR unsafe implants including implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure).
* High risk of complete AV block after TAVR, with the need of permanent pacemaker.
* Claustrophobia precluding MRI scanning.

Anatomical and CT Exclusion Criteria:

* Severe peripheral arterial, abdominal aortic, or thoracic aortic disease that precludes delivery sheath, vascular access or filter deployment.
* Presence of cardiovascular implant in aorta and/or peripheral access vessels.
* Access vessels with excessive tortuosity.
* Aortic arch, which is heavily calcified, severely atheromatous, or severely tortuous.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 30 days post procedure
  MACCE includes the composite of death, all stroke, acute kidney injury (AKI) stage 3 or 4 within 7 days post-index procedure Valve Academic Research Consortium 3 (VARC-3) and any major vascular complication (VARC-3)
Total New Lesion Volume | 8-72 hours post procedure
  Total new lesion volume (TNLV) in the brain assessed by diffusion weighted magnetic resonance images (DW-MRI)

SECONDARY OUTCOMES:
Stroke | 30 days post procedure
  Incidence of all stroke events

OTHER OUTCOMES:
Performance | During procedure
  Technical success (% of patients with successful device deployment, position and retrieval) and procedure success (% of patients with technical device success and no device-related safety events)
Mortality & Stroke Rates | 30 days post procedure
  Incidences of all-cause mortality, major stroke, minor stroke events
Freedom from Lesions | 8-72 hours post procedure
  Measure presence or absence of new lesions in the brain, assessed by diffusion weighted magnetic resonance images (DW-MRI)
Average Lesion Size | 8-72 hours post procedure
  Measure average lesion size in the brain, assessed by diffusion weighted magnetic resonance images (DW-MRI)
Neurological Outcomes-National Institute of Health Stroke Scale (NIHSS) | 30 days post procedure
  Use National Institute of Health Stroke Scale (NIHSS) to measure stroke severity on a scale of 0-41 (low score is better outcome).
Neurological Outcomes-Montreal Cognitive Assessment (MoCA) | 30 days post procedure
  Use Montreal Cognitive Assessment (MoCA) to measure cognitive impairment on a scale of 0-30 (high score is better outcome).
Neurological Outcomes-Modified Rankin Scale (MRS) | 30 days post procedure
  Use Modified Rankin Scale (MRS) to measure neurological disability on scale of 0-6 (Low score is better outcome)
Major Vascular Complication & Bleeding | During procedure
  Measure major vascular complications (as defined by VARC-3) & major bleeding (Type 3, Type 4 as defined by VARC- 3)
Hospital Readmissions | 30 days post procedure
  Measure number of hospital readmissions at 30 days and number of ICU readmissions during hospital stay and 30 days
Index Hospital Length of Stay (LOS) | Through 30 days
  Measure Index hospitalization LOS
Index Hospitalization ICU Length of Stay (LOS) | Through 30 days
  Measure Index hospitalization ICU length of stay
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 30 days post procedure
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a self-reported questionnaire that measures physical function, symptoms, social function, and quality of life, on a scale from 0 to 100 (higher score is better outcome).
Short Form (SF-12) Questionnaire | 30 days post procedure
  The Short Form (SF-12) Questionnaire is a self-reported questionnaire that assess the impact of health on an individual's everyday life, on a scale from 0 to 100 (higher score is better health).

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - NCH Baker Hospital-Naples Heart Institute, Naples, Florida
  - St. Vincent Hospital, Indianappolis, Indiana
  - Henry Ford Hospital, Detroit, Michigan
  - St. Lukes Hospital Of Kansas City, Kansas City, Missouri
  - Cumc/Nyph, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute (aka Riverside Methodist Hospital), Columbus, Ohio
  - University of Virginia Medical Center, Charlottesville, Virginia
- Australia (2):
  - St Andrews War Memorial Hospital, Spring Hill, Queensland
  - Monash Health Public, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No